CLINICAL TRIAL: NCT01975311
Title: Effect of Lumbopelvic Manipulation on Hip and Knee Neuromuscular Activity, Pain Intensity, and Functional Activity in People With Patellofemoral Pain Syndrome.
Brief Title: Effect of Lower Back Treatment in People With Patellofemoral Pain Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17284
Record Dates: First submitted 2013-10-28; First posted 2013-11-04 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2014-11

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lumbopelvic Manipulation (Experimental): Participants in this group will receive lumboplevic manipulation twice within a week.
  Interventions: Other: Lumbopelvic Manipulation
- Passive lumbar spine flexion and extension (Placebo Comparator): Participants in this group will receive passive lumbar spine flexion and extension for 1 min twice within a week.
  Interventions: Other: Passive lumbar spine flexion and extension

INTERVENTIONS:
Other: Lumbopelvic Manipulation — High-velocity low-amplitude non-specific lumbopelvic thrust manipulation
  Arms: Lumbopelvic Manipulation
Other: Passive lumbar spine flexion and extension — Passive lumbar spine flexion and extension without reaching the physiological end feel for 1 min from a side lying position.
  Arms: Passive lumbar spine flexion and extension

SUMMARY:
The purpose of this study is to determine if a lower back treatment would change the knee pain intensity and the level of functional activities as well as the muscle activities in people with anterior knee pain. The investigators hypothesized that the lower back treatment may change the hip and knee muscle activities as well as reduce the knee pain intensity and improve the functional activities in people with anterior knee pain.

ELIGIBILITY:
Inclusion Criteria:

* Insidious onset of symptoms of non-traumatic origin.
* Pain with patellar facet palpation or compression.
* anterior or retropatellar knee pain during at least two of the following activities: (a) ascending stairs, (b) descending stairs, (c) kneeling, (d) squatting, (e) hopping, (f) running, (j) jumping, (h) prolonged sitting for more than 20 minutes.

Exclusion Criteria:

* History of spine, hip or knee surgery.
* History of hip pathology or other knee condition.
* Current significant injury of any lower extremity joints.
* Pregnancy.
* Sign of nerve root compression.
* Osteoporosis or history of compression fracture.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2012-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Electromyography (EMG) of the hip and knee muscle | The EMG data will be collected within one week for all participants in both groups.
  EMG unit will be used to study the hip and knee muscle activities.

SECONDARY OUTCOMES:
Pain Visual Analog Scale (VAS) | The pain VAS data will be collected within one week for all participants in both groups
Lower Extremity Functional Scale (LEFS) | The LEFS data will be collected within one week for all participants in both groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Texas Woman's University, School of Physical Therapy - Dallas Campus, Dallas, Texas, United States